CLINICAL TRIAL: NCT00286338
Title: Comparison of Monitors of Fluid Therapy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: des.prost-1
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Hypovolemia
Keywords: Fluid therapy; Monitoring
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The investigators want to correlate different methods to guide fluid therapy. The investigators know that guidance by esophagus doppler technique has improved outcome and want to correlate other already used techniques to esophagus doppler.

DETAILED DESCRIPTION:
Fluid therapy before and under surgery can be guided by measurement of the hearts ability to eject blood (cardiac output). By doing this it has been shown that the occurrence of nausea,vomiting and complications generally can be reduced. The function of the heart has been measured with a probe in the esophagus in in earlier studies. We want to correlate these results with other techniques by which fluid therapy also is guided in daily practice. These are: SVO2, modelflow (finapres)and NIRS.

These methods are noninvasive except SVO2 measurement which requires a central venous catheter (CVK). Therefore we have chosen a population in which CVK is standard in our institution. We thereby don´t apply any further risks than daily practice and the project is considered as a quality assessment of used standards.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Elective urological surgery in which a central venous catheter is routinely administered
* Informed consent

Exclusion Criteria:

* Age 70 years or older
* No informed consent
* Pathology in the esophagus that contraindicates use off gastric tube and esophagus doppler
* ASA III or above

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-02; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, M.D., Ph.D, Study Director — dept of surgical patophysiology
Locations (1):
- Dept of anesthesia 2041, ABD centre, Rigshospitalet, Blegdamsvej, Copenhagen, Denmark